CLINICAL TRIAL: NCT05794126
Title: A Clinical Comparison of Two Soft Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C22-726 (EX-MKTG-147)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (Experimental): Participants wore Lens 1 for 15 minutes (Period 1)
  Interventions: Device: Lens 1
- Lens 2 (Experimental): Participants wore Lens 2 for 15 minutes (Period 2)
  Interventions: Device: Lens 2

INTERVENTIONS:
Device: Lens 1 — Soft multifocal hydrogel contact lens for 15 minutes
  Arms: Lens 1
Device: Lens 2 — Soft multifocal silicone hydrogel contact lens for 15 minutes.
  Arms: Lens 2

SUMMARY:
The study objective was to gather short-term clinical performance data for two soft multifocal contact lenses.

DETAILED DESCRIPTION:
The aim of this subject-masked, non-randomized, non-dispensing study was to evaluate the short-term clinical performance of a soft multifocal hydrogel contact lens when compared to a soft silicone multifocal hydrogel lens after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

1. They were at least 42 years of age and had capacity to volunteer.
2. They understood their rights as a research subject and were willing and able to sign a Statement of Informed Consent.
3. They had had a full eye examination within the past two years (by self-report).
4. They were willing and able to follow the protocol.
5. They habitually used vision correction for near vision (multifocal soft contact lenses, sphere lenses for monovision, sphere lenses for distance vision correction and spectacles for near vision correction, or had a different spectacle prescription for distance and near vision correction) and had done so for at least the past three months.
6. They had refractive astigmatism of no greater than -0.75DC.
7. They could be fitted with the study lenses within the power range available, and achieved binocular distance HCVA of +0.20 or better in the study lenses.

Exclusion Criteria:

Subjects were not eligible to take part in the study if:

1. They had an ocular disorder which would normally contra-indicate contact lens wear.
2. They had a systemic disorder which would normally contra-indicate contact lens wear.
3. They were using any topical medication such as eye drops or ointment.
4. They were aphakic.
5. They had had corneal refractive surgery.
6. They had any corneal distortion resulting from previous hard or rigid lens wear or had keratoconus.
7. They were pregnant or lactating.
8. They had an eye or health condition including an immunosuppressive or infectious disease which could, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens 1: All participants wore Lens 1 for 15 minutes (Period 1)
- Lens 2: All participants wore Lens 2 for 15 minutes (Period 2)
Period: Period 1: Lens 1, 15 Minutes
Arm/Group | Lens 1 | Lens 2
Started | 47 | 0 (All participants received Lens 1 in Period 1.)
Completed | 47 | 0
Not Completed | 0 | 0
Period: Period 2: Lens 2, 15 Minutes
Arm/Group | Lens 1 | Lens 2
Started | 0 (All participants received Lens 2 in Period 2.) | 47
Completed | 0 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes study participants that completed all study visits
Arm/Group | All Study Participants
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Score
Description: Subjective Overall Score was assessed using the 0-100 visual analogue scale where 0=Extremely poor, cannot use lenses and 100=Excellent=Highly impressed with these lenses overall
Time Frame: 15 Minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens 1: Participants that received Lens 1
- Lens 2: Participants that received Lens 2
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 47 | 47
score on a scale | 71.4 (18.0) | 80.3 (14.7)

2. Secondary Outcome: Subjective Comfort
Description: Subjective Comfort Score was assessed using the 0-100 visual analogue scale where 0=Extremely uncomfortable, causes pain, cannot be tolerated and 100=Excellent, cannot be felt
Time Frame: 15 Minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 47 | 47
score on a scale | 75.0 (20.9) | 88.9 (12.2)

3. Secondary Outcome: Subjective Vision
Description: Subjective Vision Score (distance and near) was assessed using the 0-100 visual analogue scale where 0=Unacceptable, cannot be worn and 100=Excellent, unaware of any visual loss
Time Frame: 15 Minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 47 | 47
score on a scale
  Distance Vision | 72.3 (17.1) | 78.4 (15.8)
  Near Vision | 77.4 (18.2) | 79.6 (15.7)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2.5 hours
Arm/Group | Lens 1 | Lens 2
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT05794126/Prot_SAP_000.pdf